CLINICAL TRIAL: NCT06255522
Title: Clinical and Anatomical Factors Influencing Accuracy in Fully Guided Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Professor, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REST-ECL-2023-08
Record Dates: First submitted 2023-11-22; First posted 2024-02-13 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Edentulous Mouth
Keywords: Fully guided implant placement; Accuracy
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fully guided implant placement (Experimental): Through guided surgery implant placement will be performed in maxilla or mandibula in a one stage surgery. The final position will be compare with the initial digital implant planning.
  Interventions: Procedure: Fully guided implant placement

INTERVENTIONS:
Procedure: Fully guided implant placement — Through guided surgery, previously planned and designed based on CBCT study and CAD/CAM scanning, implant placement of Conelog Progressive line implants (Biohorizons Camlog, Iberia) will be performed in maxilla or mandibula in a one stage surgery. Postoperative CBCT in ECO mode (35μSv) will be taken after the implant placement to assess the final position and comparing with the initial digital planning.

SUMMARY:
The importance of the stability of hard and soft tissues has been shown to be of paramount importance for long-term implant success. To reach optimal functional and aesthetic outcomes, implant placement must be planned accordingly to prosthetic needs and design. Prosthetically driven implant placement is based on a diagnostic prosthetic set-up that is followed by precise implant planification and placement using CBCT and intraoral scanning.

The aim of this research is to evaluate how the clinical and anatomical factors can influence the 3D position of guided surgery.

DETAILED DESCRIPTION:
After assessing the fulfillment of the inclusion criteria, pre-operative cone beam computed tomography (CBCT) (Newtom, Cefla S.C.) and intraoral digital impressions (Trios®, 3Shape Dental Systems, Denmark) will be obtained for each patient to achieve a digital wax-up and a presurgical plan for the exact position of the implants by a single calibrated operator (RP).

Every patient could have a maximum of four implants to be placed (one per quadrant), in those cases, each implant will be placed with its own surgical guide.

The digital imaging and communications in medicine (DICOM) files will be imported to a guided-surgery planning software (Codiagnostix, Dental wings) to perform an implant planning based on the digital wax up; in this step the assessment of the mucosal thickness will be performed using the STL and the DICOM files superimposed. The measurement will be taken from the crestal bone until the soft tissue surface (mm).

Furthermore, a surgical guide will be designed, and 3D printed (SprintRay Pro S; SprintRay Inc) with implant guide resin (SprintRay EU Surgical Guide Clear; SprintRay Inc) by RP for the surgical procedure, supported by the whole dental arch, and reinforced with one bar across the arch.

Through guided surgery, previously planned and designed based on CBCT study and CAD/CAM scanning, placement of Conelog Progressive line implants (Biohorizons Camlog, Iberia) will be performed in maxilla or mandibula in a one stage surgery by a 8 years' experience operator (GB).

Implant placement will be fully guided and a postoperative CBCT in ECO mode (35μSv) will be taken after the implant placement to assess the final position.

Both CBCT will be aligned (pre-op scan and post-op scan) to make calculations by a single evaluator (AB) included the following: (1) angle: angle deviation measured in degrees; (2) base: deviation at implant shoulder in millimeters; (3) tip: deviation at implant apex in millimeters; (4) 3D offset: global deviation in 3D directions in millimeters; (5) mesiodistal deviation in millimeters: (+) deviated to the distal direction and (-) deviated to the mesial direction; (6) buccolingual deviation in millimeters: direction: (+) deviated to lingual direction and (-) deviated to buccal direction; and (7) apicocoronally deviation in millimeters: direction: ( +) deviated in the apical direction. and (-) deviated in the coronal direction.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 to 60 years old.
* Periodontally stable patients. Adequate oral hygiene with less than 15% Full Mouth Plaque Score (FMPS).
* Patients who need dental implant treatment without simultaneous regeneration.
* Ability to follow instructions and availability to attend for regular compliance during the entire study.
* With presence of partial edentulism (at least 6 remaining teeth distributed in the dental arch to support the guide).

Exclusion Criteria:

* Active infections
* Untreated periodontal disease
* Heavy smokers (>10 cigarettes per day)
* Drug / Alcohol dependency
* Medical condition contraindicating implants dependency
* Patients under bisphosphonate therapy
* Limited mouth opening
* Edentulous patients or with les than 6 teeth.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of fully guided implant placement | Baseline
  Both CBCT will be aligned (pre-op scan and post-op scan) to make calculations by a single evaluator (AB) included the following: (1) angle: angle deviation measured in degrees; (2) base: deviation at implant shoulder in millimeters; (3) tip: deviation at implant apex in millimeters; (4) 3D offset: global deviation in 3D directions in millimeters; (5) mesiodistal deviation in millimeters: (+) deviated to the distal direction and (-) deviated to the mesial direction; (6) buccolingual deviation in millimeters: direction: (+) deviated to lingual direction and (-) deviated to buccal direction; and (7) apicocoronally deviation in millimeters: direction: ( +) deviated in the apical direction. and (-) deviated in the coronal direction.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Blasi Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT06255522/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT06255522/ICF_001.pdf